CLINICAL TRIAL: NCT07227805
Title: Evaluation of the Safety and Performance of the Novel Medtronic Experimental Automated Insulin Delivery System (NMX8) in People Living With Diabetes
Brief Title: Evaluation of the Safety and Performance of the Novel Medtronic Experimental Automated Insulin Delivery System (NMX8) in People Living With Diabetes (NEXUS)
Acronym: NEXUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP352
Record Dates: First submitted 2025-11-11; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Diabetes (Insulin-requiring, Type 1 or Type 2)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment arm (NMX8) (Experimental): Subjects randomized to the Treatment group will use the MiniMed™ NMX8 system
  Interventions: Device: NMX8
- Control arm (780G) (Active Comparator): Subjects randomized to the Control arm will continue to use the MiniMed™ 780G.
  Interventions: Device: 780G

INTERVENTIONS:
Device: NMX8 — Subjects will start using the MiniMed™ NMX8 system for 12 weeks
  Arms: Treatment arm (NMX8)
Device: 780G — Subjects will continue to use the MiniMed™ 780G for 12 weeks
  Arms: Control arm (780G)

SUMMARY:
This study will demonstrate the safety and performance of the Novel Medtronic Experimental Automated Insulin Delivery system named MiniMed™ NMX8 system in people living with insulin-requiring diabetes in comparison with the MiniMed™ 780G system.

DETAILED DESCRIPTION:
This study is a pre-market, interventional, prospective, open-label, multi-center and randomized controlled clinical study.

The study consists of a run-in phase and a study phase.

Run-in Phase:

The purpose of the run-in phase is to collect baseline CGM data while subjects are on 780G therapy in Auto Mode. All subjects will use the Simplera Sync sensor.

At the end of the run-in phase, subjects will be randomly allocated to one of the two study arms (Treatment arm or Control arm).

Study Phase:

During the 12-week study phase, subjects will either start using the MiniMed™ NMX8 system (Treatment arm) or will continue to use the MiniMed™ 780G in Auto Mode (Control arm). During the study phase, all subjects will use the Simplera™ Sync sensor.

ELIGIBILITY:
Inclusion Criteria:

1. Is aged ≥2 years old at time of screening.
2. Has a clinical diagnosis of Type 1 or Type 2 diabetes for ≥ 6 months prior to screening as determined via medical record by an individual qualified to make a medical diagnosis.
3. Is on MiniMed™ 780G with Simplera Sync sensor for at least 3 months before screening.
4. Has a glycosylated hemoglobin (HbA1c) <11% (97 mmol/mol) at time of screening visit as processed at Point of Care (PoC) or local lab.
5. Must have a minimum daily insulin requirement (Total Daily Dose) of ≥ 6 units and a maximum of 250 units
6. Willing to switch to approved insulin per insulin pump labeling.
7. Investigator has confidence that the subject, parent(s)/legal guardian(s) can successfully operate all study devices and is capable of adhering to study visit schedule per protocol.
8. Subject, Parent(s)/legal guardian(s) is willing to participate in all training sessions as directed by study staff.
9. Subject, Parent(s)/legal guardian(s) is willing and able to provide written informed consent.
10. For subject with Type 2 Diabetes only: Is on stable dose of anti-diabetic medication (other than insulin) (e.g., pramlintide, DPP-4 inhibitor, GLP-1 and GIP agonists/mimetics, metformin, SGLT2 inhibitors) for the last 3 months prior to screening. NB: Subject should not change type or dose of medication during the course of the study.
11. For Israel only: Subject, Parents(s)/legal guardian(s) is fluent in English.

Exclusion Criteria:

1. Has Addison's disease, growth hormone deficiency, hypopituitarism or definite gastroparesis, uncontrolled coeliac disease, uncontrolled thyroid disorder, or poorly controlled asthma, per investigator judgment.
2. For subjects with Type 1 Diabetes only: Is using any anti-diabetic medication other than insulin 6 months before screening or plan on using during the study (e.g., pramlintide, DPP-4 inhibitor, GLP-1 and GIP agonists/mimetics, metformin, SGLT2 inhibitors).
3. Has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any chronically oral, injectable, or IV glucocorticoids during the course of the study, per investigator judgement
4. Has had renal failure defined by creatinine clearance <30 ml/min, as assessed by local lab test ≤ 6 months before screening or performed at screening at local lab, as defined by the creatinine-based Cockcroft, CKD-EPI or MDRD equations.
5. Has active or severe retinopathy in the last 6 months before screening
6. Has any unresolved adverse skin conditions in the area of sensor placement (e.g. psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
7. Has any other disease or condition that may preclude the patient from participating in the study, per investigator judgment.
8. History of 2 or more DKA events in the last 3 months before screening.
9. Has had Hyperosmolar Hyperglycemic State (HHS) in the last 6 months before screening.
10. Is using hydroxyurea at time of screening or plans to use it during the study
11. Women of child-bearing potential who have a positive pregnancy test at screening or plan to become pregnant during the course of the study.
12. Women who are breastfeeding.
13. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or device in the last 2 weeks before screening, as per investigator judgment.
14. Subject is currently abusing illicit drugs, marijuana, alcohol or prescription drugs (other than nicotine), per investigator judgment.
15. Subject, Parent(s)/legal guardian(s) are part of research staff involved with the study.
16. Subject, Parent(s)/legal guardian (s) are legally incompetent, illiterate, or vulnerable.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2027-03-17 (Estimated); Study Completion 2027-03-17 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | During the 12-week study phase
  The between-treatment (control arm with 780G system versus treatment arm with NMX8 system) difference during the study phase in the percentage of time that the sensor glucose measurement is in the target range, 70 to 180 mg/dL (3.9-10.0 mmol/L) with a non-inferiority testing.

SECONDARY OUTCOMES:
Secondary Endpoint 1 | End of 12-week Study Phase
  The between-treatment (NMX8 system arm versus 780Gm system arm) difference in HbA1c (%) at the end of the 3-month study phase with a non-inferiority testing.
Secondary endpoint 2 | During the 12-week Study Phase
  The between-treatment (NMX8 system arm versus 780Gm system arm) difference in % of Time spent in target range (70 to 180 mg/dL [3.9 - 10.0 mmol/L]) during the study phase with superiority test.
Secondary Endpoint 3 | End of the 12-week Study Phase
  The between-treatment (NMX8 system arm versus 780Gm system arm) difference in HbA1c (%) at the end of the 3-month study phase with superiority testing.

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Ohad Cohen, MD, Study Chair — Medtronic Diabetes

IPD SHARING:
Plan to Share IPD: No